CLINICAL TRIAL: NCT03777345
Title: Evaluation of Periodontal Health of the Abutment Teeth in Partial Dentures Made of Injection Molded PEEK Framework Versus Cobalt Chromium Framework in Mandibular Kennedy Class I Edentulous Cases
Brief Title: Comparison Between Injection Molded Polyetheretherketone (PEEK) Framework and Cobalt Chromium Framework Removable Partial Dentures Regarding Periodontal Health of Abutment Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hefny Zidan, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-11-28
Record Dates: First submitted 2018-12-11; First posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Mandibular Prosthesis User

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cobalt-chromium framework partial dentures (Active Comparator): It's the gold standard biocompatible metal alloy used in thin sections, provide high strength and stiffness ,conduct heat and cold for a more natural experience, and is resistant to corrosion but their disadvantages include esthetic issues with metal display, oral galvanism, adverse tissue reactions,and osteolysis of abutment teeth.
  Interventions: Device: cobalt-chromium framework partial dentures
- PEEK framework partial dentures (Experimental): It's a promising polymer-based framework has recently been introduced which is made of polyetheretherketone polymer frame combined with acrylic resin denture teeth and a conventional acrylic resin denture base.
  Interventions: Device: PEEK framework partial dentures

INTERVENTIONS:
Device: cobalt-chromium framework partial dentures — It's a biocompatible metal alloy used in thin sections and are less bulky, provide high strength and stiffness ,conduct heat and cold for a more natural experience, enable designs that minimize the covering of the gingival margins, allow for a stable denture base, and is resistant to corrosion. Disadvantages include hypersensitivity, esthetic issues with metal display, oral galvanism, adverse tissue reactions, osteolysis of abutment teeth, and biofilm production .
  Arms: cobalt-chromium framework partial dentures
Device: PEEK framework partial dentures — It's a promising polymer-based framework material has recently been introduced which is made of polyetheretherketone polymer frame combined with acrylic resin denture teeth and a conventional acrylic resin denture base.
  Arms: PEEK framework partial dentures

SUMMARY:
This study is aiming to evaluate the periodontal status of the abutment teeth in Polyetheretherketone ( PEEK ) framework partial dentures compared with cobalt-chromium ones in mandibular kennedy class I edentulous cases aiming to preserve the optimum periodontal health of the abutment teeth .

ELIGIBILITY:
Inclusion Criteria:

* Kennedy Class I partially edentulous subjects indicated for framework partial denture

Exclusion Criteria:

* 1- uncooperative patients . 2- bad oral hygiene patients .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Periodontal status | Change in periodontal status will be assessed at base line , after one month and after 3 months .
  periodontal status of the abutment teeth assessed by a periodontal chart .

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abdel-Bary SK, Rostom EM, Elboarey AN. Thermoplastic Removable Partial Dentures versus Metal Cobalt-Chromium. RESEARCH JOURNAL OF PHARMACEUTICAL BIOLOGICAL AND CHEMICAL SCIENCES. 2016 Jul 1;7(4):464-70.